CLINICAL TRIAL: NCT05717309
Title: Trajectories of Chronic Multimorbidity Patterns in Patients >65 Years Old. MTOP
Brief Title: Trajectories of Chronic Multimorbidity Patterns in Older Patients
Acronym: MTOP
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Department of Health, Generalitat de Catalunya (Other Government)
Responsible Party: Principal Investigator, Marina Lleal Custey, Principal Investigator, Corporacion Parc Tauli
Other Study IDs: CIR2021038
Record Dates: First submitted 2023-01-25; First posted 2023-02-08 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Chronic Disease
Keywords: Multimorbidity; Cluster analysis; Trajectories; Older patient; COVID-19
MeSH Terms: conditions — Chronic Disease; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Following the MRisk-COVID project, MTOP (Multimorbidity Trajectories in Older Patients) study was developed. It is a retrospective observational study using Real World Data that aims to identify patterns of chronic multimorbidity in patients aged ≥65 years and their evolution and trajectories in the previous 10 years. The secondary objective is to identify the relationship between the trajectories of multimorbidity patterns in the previous 10 years and the severity of the infection by COVID-19.

DETAILED DESCRIPTION:
Multimorbidity is associated with negative results and presents difficulties in clinical management. Recently, new methodologies are emerging based on the hypothesis that chronic conditions are associated in a non-random way forming multimorbidity patterns. However, there are few studies that study the temporal evolution and trajectories of these multimorbidity patterns, which could be associated with different prognoses and could allow better forecasting and planning. The primary objective of this analysis is to identify patterns of chronic multimorbidity in patients aged ≥65 years and their evolution and trajectories in the previous 10 years, using part of the MRisk-COVID project data. As a secondary objective, the investigators want to identify the relationship between the trajectories of multimorbidity patterns in the previous 10 years and the severity of the COVID-19 infection. This retrospective observational study has a historical cohort of 3958 patients ≥65 years of age suspected and confirmed of COVID-19 infection from February 1 to June 15, 2020 in the reference area of Parc Taulí University Hospital. The available data (real-world data) are socio-demographic and diagnostic variables provided by the Data Analytics Program for Research and Innovation in Health (PADRIS), which include sex, age and primary care diagnoses. To identify patterns of multimorbidity, the Clinical Classification Software, Chronic Condition Indicator, multiple correspondence analysis and cluster analysis using the fuzzy c-means algorithm will be used. Then, a clinical consensus process (Delphi-like) will be made of the clusters obtained. To identify the most probable trajectories along the three time points, each patient will be assigned to the cluster with the highest probability of membership. Descriptive and bivariate statistics will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Positive results of COVID-19 laboratory tests
* COVID-19 related clinical profile verified by healthcare professionals

Exclusion Criteria:

* Males >90 years (re-identification risk)

Ages: 65 Years to 94 Years | Sex: All
Age Groups: Older Adult
Study Population: Confirmed or suspected COVID-19 patients from the first wave of the pandemic, aged 65 years and over, residing in a healthcare region of about 400.000 inhabitants in a Northeast region of Spain (Vallès Occidental Est, Catalonia, Spain).
Sampling Method: Non-Probability Sample
Enrollment: 3988 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Chronic multimorbidity patterns - Time Frame 1 | Baseline (2020)
  Obtained using fuzzy c-means cluster analysis
Chronic multimorbidity patterns - Time Frame 2 | 5 years before (2015)
  Obtained using fuzzy c-means cluster analysis
Chronic multimorbidity patterns - Time Frame 3 | 10 years before (2010)
  Obtained using fuzzy c-means cluster analysis
Trajectories of chronic multimorbidity patterns | Change over 10 years
  Obtained by assigning the highest probable cluster at each time point

SECONDARY OUTCOMES:
Severe COVID-19 infection | From 27-February-2020 to 15-June-2020
  Severe COVID-19 infection was defined as the occurrence of at least one of the following conditions during any of the registered COVID-19 episodes: severe respiratory affection (including insufficiency, failure, or distress); use of respiratory support (including mechanical ventilation or oxygen therapy); septic shock; multiple organ failure (the combination of respiratory failure and any other organ failure); inflammatory response; admission to intensive care unit; and mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Corporacio Parc Taulí, Sabadell, Barcelona, Spain

REFERENCES:
- [Derived] Lleal M, Bare M, Herranz S, Orus J, Comet R, Jordana R, Bare M. Trajectories of chronic multimorbidity patterns in older patients: MTOP study. BMC Geriatr. 2024 May 30;24(1):475. doi: 10.1186/s12877-024-04925-2. PMID 38816787